CLINICAL TRIAL: NCT04797962
Title: Linkage Navigation to Enhance Initiation and Engagement in Treatment for Opioid Use Disorder to Prevent Overdose
Brief Title: Connection, Navigation, Engagement in Care and Treatment for Opioid Use Disorder
Acronym: ConNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alia Al-Tayyib, Associate Research Scientist, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-2236; R01CE00300 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): dedicated case management
  Interventions: Behavioral: Case management
- Usual care (No Intervention): usual care

INTERVENTIONS:
Behavioral: Case management — dedicated case management to address social support needs
  Arms: Intervention

SUMMARY:
The overarching goal of the study is to develop, pilot, and evaluate an intervention that aims to retain patients who initiate buprenorphine at Denver Health in ongoing treatment for opioid use disorder.

DETAILED DESCRIPTION:
Initiating patients identified with opioid use disorder in hospital settings onto buprenorphine is a relatively new strategy to prevent overdose. While the literature is beginning to amass showing the effectiveness of this strategy for initiating people into treatment, a dearth of data to describe how well people are maintained in treatment remains. The current research project aims to 1) develop an intervention to enhance engagement and retention in treatment for individuals with opioid use disorder who initiate buprenorphine at Denver Health and 2) assess acceptability, feasibility, and initial efficacy of an intervention to enhance engagement and retention in treatment for individuals with opioid disorder compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* inducted onto buprenorphine at Denver Health
* successfully completed an intake visit at Denver Health's Outpatient Behavioral Health Services clinic.

Exclusion Criteria:

* unable to provide informed consent
* unable to provide detailed contact information
* previously enrolled in the current study
* pregnant women will be excluded given that they are a priority treatment population and receive special services

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Retention in treatment at 90 days | 90 days from treatment initiation
  Defined by proportion of participants retained in care at 90 days, as measured by the total number of intakes where patient has continued to be engaged in medication assisted treatment at 90 days from start of treatment divided by the total number of intakes where patients linked to follow up dosing or prescription, for each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Alia Al-Tayyib, PhD, Principal Investigator — Denver Health
Locations (1):
- Denver Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided